CLINICAL TRIAL: NCT01306695
Title: Comparative Effectiveness of the NYU Caregiver Intervention in Latinos in Northern Manhattan
Brief Title: Northern Manhattan Caregiver Intervention Project
Acronym: NOCIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, José A. Luchsinger, Associate Professor of Medicine and Epidemiology, Columbia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAI0022; P60MD000206 (NIH)
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Dementia
Keywords: Dementia; Depressive symptoms; Caregiver Burden; Hispanic; Latino; Intervention; Geriatric Depression Scale; Zarit Caregiver Burden Scale
MeSH Terms: conditions — Dementia; Depression; Caregiver Burden | interventions — Community Health Workers; Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NYUCI (Experimental): New York University Caregiver Intervention (NYUCI) in addition to community-based case management using community health workers: The first component consists of two individual and four family counseling sessions that include relatives suggested by the caregiver.
  Interventions: Behavioral: New York University Caregiver Intervention (NYUCI)
- CHW Intervention (Other): Community-based case management using community health workers (CHWs): The CHW intervention will consist of 2 visits in month 1, followed by monthly visits until month 6.
  Interventions: Other: Community Health Worker (CHW) Case Management

INTERVENTIONS:
Behavioral: New York University Caregiver Intervention (NYUCI) — The NYU Caregiver Intervention (NYUCI) has substantial evidence of efficacy. This intervention is unique in its emphasis on family support and in providing ongoing availability of the counselor. While the NYUCI is being implemented in several communities, its effectiveness in the Hispanic community of Northern Manhattan has not been tested. The first component of the intervention consists of two individual and four family counseling sessions that include relatives suggested by the caregiver. The second component of the intervention is participation in a support group to provide the caregiver with continuous emotional support and education. The third component of the treatment is "ad hoc" counseling the continuous availability of counselors to caregivers and families to help them deal with crises and with the changing nature and severity of their relatives' symptoms over the course of the disease.
  Other Names: NYU Caregiver Intervention
  Arms: NYUCI
Other: Community Health Worker (CHW) Case Management — The CHW intervention will consist of 2 visits in month 1, followed by monthly visits until month 6. The main role of the CHW will be to provide access to existing education and referral resources about dementia and caregiving. The CHW will carry a blackberry or iPhone type device with real time access to email, text, the internet, and telephone. Thus, the CHW will be able to provide participants with real time information from pertinent websites such as CUMC, Alianza, and the NY chapter of the Alzheimer's Association. CHW will also provide participants with their phone number and email address for ad-hoc contacts.
  Other Names: CHW
  Arms: CHW Intervention

SUMMARY:
Elderly Hispanics have a higher burden of dementia compared to Non-Hispanic Whites. Furthermore, Hispanic caregivers tend to have a higher burden of care for their relatives with dementia. The objective of this project is to conduct a randomized trial in 160 Hispanic relative caregivers of persons with dementia comparing the effectiveness of New York University Caregiver Intervention to a case management intervention lead by community health workers(CHW). This trial will last 6 months. The main outcomes in the trial will be changes in depressive symptoms measured with the Geriatric Depression Scale and caregiver burden measured with the Zarit Caregiver Burden Scale. This research project will be conducted by the Northern Manhattan Center of Excellence in Comparative Effectiveness Research for Eliminating Disparities (NOCERED) funded by the National Institute on Minority Health and Health Disparities.

DETAILED DESCRIPTION:
The goal of this study is to compare the effectiveness of an existing evidence-based dementia family caregiver intervention, the New York University Caregiver Intervention (NYUCI), to community-based case management using community health workers (CHWs) in Hispanic caregivers in Northern Manhattan. The investigators will randomize 160 relative caregivers of persons with dementia to case management alone or NYUCI in addition to case management. The total duration of followup will be 6 months. We will call this project the Northern Manhattan Caregiver Intervention Project (NOCIP).

The primary aim is to compare changes from baseline to 6 months in caregiver depressive symptoms, measured with the geriatric depression scale (GDS), and in caregiver burden using the Zarit caregiver burden interview (ZBI), between the randomization arms using an Intent to treat approach. The investigators hypothesize that depressive symptoms and caregiver burden will improve or deteriorate less in the NYUCI arm compared to the case management arm at 6 months.

This project addresses one of the priority areas for comparative effectiveness research (CER) from the Institute of Medicine, "interventions for caregivers of persons with dementia". It also addresses 2 priority conditions from the Agency for Health Care Research and Quality (AHRQ): Dementia and Depression. Dementia caregiver burden is a major source of disparities in Northern Manhattan. The prevalence of dementia in Hispanics is twice that of Non-Hispanic Whites. In addition, Hispanic families tend to be reluctant to delegate the care of their relatives with dementia and consider it a family affair. Thus, the burden of care-giving for persons with dementia is much higher in Hispanic families. NOCIP will be the first study to test the effectiveness of an existing caregiver intervention, the New York University Caregiver Intervention, in the Hispanic community of Northern Manhattan. In addition, the NYUCI has been tested in spouse caregivers, and NOCIP will be the first randomized clinical trial to include non-spouse caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Must be caring for a relative with a clinical diagnosis of dementia and have the primary responsibility for their care. All people with dementia must be living at home with their caregiver when they enroll in the study.
* In each family, the person with dementia or the caregiver has to have at least one relative living in the New York City metropolitan area.
* The caregiver must be emotionally and physically capable of participating. Caregivers with clinical depression or other serious mental illness will be referred.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2011-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in Caregiver Depressive Symptoms | Up to 6 months from study completion
  Measured with the geriatric depression scale (GDS)

SECONDARY OUTCOMES:
Change in Caregiver Burden | Up to 6 months from study completion
  Measured with the Zarit Caregiver Burden Interview.

CONTACTS AND LOCATIONS:
Overall Officials: Jose Luchsinger, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Luchsinger J, Mittelman M, Mejia M, Silver S, Lucero RJ, Ramirez M, Kong J, Teresi JA. The Northern Manhattan Caregiver Intervention Project: a randomised trial testing the effectiveness of a dementia caregiver intervention in Hispanics in New York City. BMJ Open. 2012 Sep 14;2(5):e001941. doi: 10.1136/bmjopen-2012-001941. Print 2012. PMID 22983877
- [Background] Andrieu S, Aboderin I, Baeyens JP, Beard J, Benetos A, Berrut G, Brainin M, Cha HB, Chen LK, Du P, Forette B, Forette F, Franco A, Fratiglioni L, Gillette-Guyonnet S, Gold G, Gomez F, Guimaraes R, Gustafson D, Khachaturian A, Luchsinger J, Mangialasche F, Mathiex-Fortunet H, Michel JP, Richard E, Schneider LS, Solomon A, Vellas B. IAGG workshop: health promotion program on prevention of late onset dementia. J Nutr Health Aging. 2011 Aug;15(7):562-75. doi: 10.1007/s12603-011-0142-1. PMID 21808935
- [Background] Luchsinger JA, Tipiani D, Torres-Patino G, Silver S, Eimicke JP, Ramirez M, Teresi J, Mittelman M. Characteristics and mental health of Hispanic dementia caregivers in New York City. Am J Alzheimers Dis Other Demen. 2015 Sep;30(6):584-90. doi: 10.1177/1533317514568340. Epub 2015 Jan 29. PMID 25635108